CLINICAL TRIAL: NCT02012166
Title: A Double-Blind, Randomized, Placebo-Controlled, Single-Dose, 3-Period, 4 Treatment Incomplete Crossover Study to Assess the Effects of Single Oral Doses of L-001241689 on Glucagon-Induced Glycemic Excursion in Healthy Male Subjects Following Intravenous Administration of Glucagon, Sandostatine® and Insulin
Brief Title: A Study of MK-0893 on Glucagon-Induced Glycemic Excursion in Healthy Male Participants Following Intravenous Administration of Glucagon, Sandostatine® and Insulin (MK-0893-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0893-002; 2005-002198-57 (EudraCT Number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-16 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Therapeutic Uses; Pharmacologic Actions; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — N-((4-(1-(3-(3,5-dichlorophenyl)-5-(6-methoxynaphthalen-2-yl)-1H-pyrazol-1-yl)ethyl)phenyl)carbonyl)-beta-alanine; Octreotide; Insulin; Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- MK-0893 40 mg→MK-0893 200 mg→placebo (Experimental): In Part 1 of the study, participants receive MK-0893 (10 mg, 40 mg or 200 mg) or placebo on Day 1 of each period, and Sandostatine® (30 ng/kg/min), insulin (0.10 mIU/kg/min), and glucagon (3 ng/kg/min) at 24 and 72 hours post dose. In Part 2 of the study, participants receive MK-0893 (200 mg or 1000 mg) or placebo on Day 1 of each period and Sandostatine®, insulin, and glucagon at 120 hours post dose. There will be at least 21 days between administrations of study drugs.
  Interventions: Drug: MK-0893 40 mg; Drug: MK-0893 200 mg; Drug: Placebo; Biological: Sandostatine®; Biological: Insulin; Biological: Glucagon
- MK-0893 200 mg→placebo→MK-0893 10 mg (Experimental): In Part 1 of the study, participants receive MK-0893 (10 mg, 40 mg or 200 mg) or placebo on Day 1 of each period, and Sandostatine® (30 ng/kg/min), insulin (0.10 mIU/kg/min), and glucagon (3 ng/kg/min) at 24 and 72 hours post dose. In Part 2 of the study, participants receive MK-0893 (200 mg or 1000 mg) or placebo on Day 1 of each period and Sandostatine®, insulin, and glucagon at 120 hours post dose. There will be at least 21 days between administrations of study drugs.
  Interventions: Drug: MK-0893 10 mg; Drug: MK-0893 200 mg; Drug: Placebo; Biological: Sandostatine®; Biological: Insulin; Biological: Glucagon
- Placebo→MK-0893 10 mg→MK-0893 40 mg (Experimental): In Part 1 of the study, participants receive MK-0893 (10 mg, 40 mg or 200 mg) or placebo on Day 1 of each period, and Sandostatine® (30 ng/kg/min), insulin (0.10 mIU/kg/min), and glucagon (3 ng/kg/min) at 24 and 72 hours post dose. In Part 2 of the study, participants receive MK-0893 (200 mg or 1000 mg) or placebo on Day 1 of each period and Sandostatine®, insulin, and glucagon at 120 hours post dose. There will be at least 21 days between administrations of study drugs.
  Interventions: Drug: MK-0893 10 mg; Drug: MK-0893 40 mg; Drug: Placebo; Biological: Sandostatine®; Biological: Insulin; Biological: Glucagon
- MK-0893 10 mg→MK-0893 40 mg→MK-0893 200 mg (Experimental): In Part 1 of the study, participants receive MK-0893 (10 mg, 40 mg or 200 mg) or placebo on Day 1 of each period, and Sandostatine® (30 ng/kg/min), insulin (0.10 mIU/kg/min), and glucagon (3 ng/kg/min) at 24 and 72 hours post dose. In Part 2 of the study, participants receive MK-0893 (200 mg or 1000 mg) or placebo on Day 1 of each period and Sandostatine®, insulin, and glucagon at 120 hours post dose. There will be at least 21 days between administrations of study drugs.
  Interventions: Drug: MK-0893 10 mg; Drug: MK-0893 40 mg; Drug: MK-0893 200 mg; Biological: Sandostatine®; Biological: Insulin; Biological: Glucagon
- Placebo→MK-0893 1000 mg→MK-0893 200 mg (Experimental): In Part 1 of the study, participants receive MK-0893 (10 mg, 40 mg or 200 mg) or placebo on Day 1 of each period, and Sandostatine® (30 ng/kg/min), insulin (0.10 mIU/kg/min), and glucagon (3 ng/kg/min) at 24 and 72 hours post dose. In Part 2 of the study, participants receive MK-0893 (200 mg or 1000 mg) or placebo on Day 1 of each period and Sandostatine®, insulin, and glucagon at 120 hours post dose. There will be at least 21 days between administrations of study drugs.
  Interventions: Drug: MK-0893 200 mg; Drug: MK-0893 1000 mg; Drug: Placebo; Biological: Sandostatine®; Biological: Insulin; Biological: Glucagon
- MK-0893 200 mg→placebo→MK-0893 1000 mg (Experimental): In Part 1 of the study, participants receive MK-0893 (10 mg, 40 mg or 200 mg) or placebo on Day 1 of each period, and Sandostatine® (30 ng/kg/min), insulin (0.10 mIU/kg/min), and glucagon (3 ng/kg/min) at 24 and 72 hours post dose. In Part 2 of the study, participants receive MK-0893 (200 mg or 1000 mg) or placebo on Day 1 of each period and Sandostatine®, insulin, and glucagon at 120 hours post dose. There will be at least 21 days between administrations of study drugs.
  Interventions: Drug: MK-0893 200 mg; Drug: MK-0893 1000 mg; Drug: Placebo; Biological: Sandostatine®; Biological: Insulin; Biological: Glucagon
- MK-0893 1000 mg→MK-0893 200 mg→placebo (Experimental): In Part 1 of the study, participants receive MK-0893 (10 mg, 40 mg or 200 mg) or placebo on Day 1 of each period, and Sandostatine® (30 ng/kg/min), insulin (0.10 mIU/kg/min), and glucagon (3 ng/kg/min) at 24 and 72 hours post dose. In Part 2 of the study, participants receive MK-0893 (200 mg or 1000 mg) or placebo on Day 1 of each period and Sandostatine®, insulin, and glucagon at 120 hours post dose. There will be at least 21 days between administrations of study drugs.
  Interventions: Drug: MK-0893 200 mg; Drug: MK-0893 1000 mg; Drug: Placebo; Biological: Sandostatine®; Biological: Insulin; Biological: Glucagon

INTERVENTIONS:
Drug: MK-0893 10 mg — MK-0893 10 mg administered orally in 240 mL of water
  Arms: MK-0893 10 mg→MK-0893 40 mg→MK-0893 200 mg; MK-0893 200 mg→placebo→MK-0893 10 mg; Placebo→MK-0893 10 mg→MK-0893 40 mg
Drug: MK-0893 40 mg — MK-0893 40 mg administered orally in 240 mL of water
  Arms: MK-0893 10 mg→MK-0893 40 mg→MK-0893 200 mg; MK-0893 40 mg→MK-0893 200 mg→placebo; Placebo→MK-0893 10 mg→MK-0893 40 mg
Drug: MK-0893 200 mg — MK-0893 200 mg administered orally in 240 mL of water
  Arms: MK-0893 10 mg→MK-0893 40 mg→MK-0893 200 mg; MK-0893 1000 mg→MK-0893 200 mg→placebo; MK-0893 200 mg→placebo→MK-0893 10 mg; MK-0893 200 mg→placebo→MK-0893 1000 mg; MK-0893 40 mg→MK-0893 200 mg→placebo; Placebo→MK-0893 1000 mg→MK-0893 200 mg
Drug: MK-0893 1000 mg — MK-0893 1000 mg administered orally in 240 mL of water
  Arms: MK-0893 1000 mg→MK-0893 200 mg→placebo; MK-0893 200 mg→placebo→MK-0893 1000 mg; Placebo→MK-0893 1000 mg→MK-0893 200 mg
Drug: Placebo — Placebo administered orally in 240 mL of water
  Arms: MK-0893 1000 mg→MK-0893 200 mg→placebo; MK-0893 200 mg→placebo→MK-0893 10 mg; MK-0893 200 mg→placebo→MK-0893 1000 mg; MK-0893 40 mg→MK-0893 200 mg→placebo; Placebo→MK-0893 10 mg→MK-0893 40 mg; Placebo→MK-0893 1000 mg→MK-0893 200 mg
Biological: Sandostatine® — Sandostatine® is a somatostatin analogue. At 24 and at 72 (Part I) or 120 (Part II) hours postdose, simultaneous infusions of the Sandostatine®, insulin, and glucagon will be administered over a 2-hour period. These compounds are IV compatible and will be combined in one syringe. Intravenous Sandostatine® will be administered at 30 ng/kg/min.
  Other Names: Octreotide acetate
Biological: Insulin — At 24 and at 72 (Part I) or 120 (Part II) hours postdose, simultaneous infusions of the Sandostatine®, insulin, and glucagon will be administered over a 2-hour period. These compounds are IV compatible and will be combined in one syringe. Intravenous insulin will be administered at 0.10 milli-international unit (mIU)/kg/min.
  Other Names: Humuline Regular, Insulin for human injection
Biological: Glucagon — At 24 and at 72 (Part I) or 120 (Part II) hours postdose, simultaneous infusions of the Sandostatine®, insulin, and glucagon will be administered over a 2-hour period. These compounds are IV compatible and will be combined in one syringe. Intravenous glucagon will be administered at 3 ng/kg/min.
  Other Names: Glucagen

SUMMARY:
This is a study to assess the pharmacokinetics, safety, and tolerability of sequential single oral doses of MK-8093 10 mg, 40 mg, 200 mg, or placebo to MK-8093 (Part 1) depending on treatment assignment in young healthy male participants. In Part 2 of this study, sequential single oral doses of MK-8093 200 mg, 1000 mg or placebo to MK-8093 depending on treatment assignment will be evaluated. The primary hypothesis of the study is that at least one dose of MK-0893 will produce greater reduction of glucagon-induced glycemia as compared to placebo following the infusion of glucagon, Sandostatine®, and basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Body Mass Index of between 18 and 28 kg/m^2, or up to 30 kg/m^2 with approval of sponsor
* Non-smoker for at least 6 months
* Willing to avoid strenuous physical activity
* Willing to avoid alcohol, caffeine, and grapefruit juice consumption

Exclusion Criteria:

* History of renal, neurologic, gastrointestinal or respiratory disease or any gastrointestinal surgery
* History of multiple and/or severe allergies to a prescription, nonprescription or investigational drug or food
* History of any cardiovascular/cardiac disease
* History of any hepatic disease and primary biliary cirrhosis
* History of hypoglycemia or glucose intolerance, type 1 diabetes, or type 2 diabetes
* Requires or anticipates use of prescription or nonprescription medications, including herbal remedies
* A user of any illicit drugs or a history of drug or alcohol abuse
* Surgery, donated a unit of blood, or participated in another clinical study within 4 weeks prior to study participation
* History of hypersensitivity to insulin, glucagon, or Sandostatine®.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Post-infusion Incremental Glucose Area Under the Plasma Concentration Versus Time Curve [AUC0-240 min] Study Part 1 | Up to 76 hours postdose
Post-infusion Incremental Glucose Area Under the Plasma Concentration Versus Time Curve [AUC0-240 min] Study Part 2 | Up to 124 hours postdose

SECONDARY OUTCOMES:
Number of Participants With An Adverse Event (AE) | Up to 12 weeks
Number of Participants Who Discontinued Study Treatment Due To AEs | Up to 21 days of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC